CLINICAL TRIAL: NCT05946577
Title: Association Between Tinnitus and Hearing Loss in Patients With Locally Advanced Head and Neck Cancer Treated by Concomitant Chemoradiotherapy or Exclusive Radiotherapy: a Prospective and Multicenter Study
Brief Title: Association Between Tinnitus and Hearing Loss in Locally Advanced Head and Neck Cancer Treated by Radiotherapy Alone or With Chemotherapy: a Prospective and Multicenter Study
Acronym: AURACCO
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230058; IDRCB 2022-A02685-38 (Other: ANSM)
Record Dates: First submitted 2023-05-05; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Head Cancer; Neck Cancer
Keywords: Head and neck cancer; HNSCC; Undifferentiated nasopharyngeal cancer; UCNT; Salivary gland cancer; Radiotherapy; Chemoradiotherapy; Radiochemotherapy; Chemotherapy; Cisplatin; Ototoxicity; Tinnitus; Hearing loss
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms; Ototoxicity; Tinnitus; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated by chemoradiotherapy with high dose of cisplatin: radiotherapy 60-70 Gy in 30-35 fractions with concomitant chemotherapy by cisplatin 100 mg/m2 every 3 weeks (week 1, 3 and 7)
- Patients treated with exclusive radiotherapy or radiotherapy with non-ototoxic chemotherapy: patient ineligible for chemotherapy with cisplatin:
  * exclusive radiotherapy: 60-70 Gy in 30-35 fractions
  * radiotherapy with a non-ototoxic chemotherapy (due to contraindication to cisplatin): 60-70 Gy in 30-35 fractions

SUMMARY:
The aim of the AURACCO study is to evaluate the association between the onset of tinnitus and hearing loss in patients with locally advanced head and neck cancer treated by concomitant chemoradiotherapy or exclusive radiotherapy

DETAILED DESCRIPTION:
Radiotherapy with or without concomitant chemotherapy is the standard of care for patients diagnosed with locally advanced head and neck cancer.

This treatment is associated with many side effects, especially tinnitus and hearing loss affecting patients' quality of life. Theses toxicities are due to chemotherapy and radiotherapy, with a synergic effect.

The effects of chemoradiotherapy on hearing loss are already well documented but very limited data are available on the onset of tinnitus.

Currently, no study established a correlation between tinnitus and hearing loss after treatment by chemoradiotherapy or exclusive radiotherapy. The main question we aim to answer is whether the development of tinnitus during treatment can be a precursor to hearing loss?

Clinical data will be collected prospectively in 4 centers in Paris (Hôpital Tenon, Hôpital La Pitié-Salpêtrrière, Hôpital Saint-Louis and Hôpital Européen Georges Pompidou) to collect :

* Patient data :
* Birth date (age at diagnosis)
* Tobacco use (active : yes/no, quantity in pack-year)
* Alcohol use (active : yes/no, quantity in g/day)
* Sex
* Disease data :
* Primitive site (oral cavity, nasopharynx, oropharynx, larynx, sinus, salivary gland, carcinoma with unknown primitive)
* Histological type
* HPV status
* TNM stage
* Data at diagnosis
* Treatment data :
* Post-operative situation (yes/no)
* Radiotherapy dose received and number of fraction
* Mean and max doses received in Gy on the right and left cochleas
* Other otototoxic treatment taken during radiotherapy
* Evaluation data :
* Tinnitus evaluation (using SOMA-LENT criteria)
* Audiogram with measures at 0,25, 0,5,

  1, 2, 4, 6, 8, 10 and 12,5 kHz
* Check for hearing "microloss"
* If tinnitus present : acouphénométrie
* If hearing aid fitting indication : APHAB (Abbreviated Profile of Hearing Aid Benefit) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patient with locally advanced or post-operative ENT cancer with high risk of recurrence
* Patient ≥ 18 years
* Absence of prior chemotherapy or radiotherapy
* Patient eligible for chemotherapy with cisplatin according to the standard regimen: radiotherapy delivering 60-70 Gy in 30-35 fractions spread over 6 to 7 weeks associated with chemotherapy with cisplatin 100 mg/m2 every 3 weeks (i.e. at week 1, 4 and 7)
* Patient ineligible for cisplatin chemotherapy receiving:

  * Either exclusive radiotherapy (age > 70 years, contraindication: renal failure, patient wearing a device): radiotherapy delivering 60-70 Gy in 30-35 fractions spread over 6 to 7 weeks.
  * either chemoradiotherapy with a chemotherapy protocol different from the standard scheme (due to a contraindication to cisplatin): radiotherapy delivering 60-70 Gy in 30-35 fractions spread over 6 to 7 weeks associated with non-standard chemotherapy ototoxic (cetuximab or carboplatin-5FU)

Exclusion Criteria:

* Tinnitus grade ≥ 2 according to the SOMA-LENT scale
* Patient fitted for hearing disorders
* Significant cognitive disorders that may compromise the performance of the various assessments
* Patients treated with weekly cisplatin
* Patient's refusal to participate in research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients followed in Hôpital Tenon, Hôpital Pitié-Salpétrière, Hôpital Saint-Louis or Hôpital Européen Georges Pompidou for a histological diagnosis of locally advanced head and neck cancer with an indication for concomitant chemoradiotherapy or exclusive radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Association between the onset of tinnitus and hearing loss at 3 months after treatment | 3 months after treatment
  Evaluation of the tinnitus on each ear. Hearing loss is defined as a loss of more than 20 dB compared to the measurement made at inclusion

SECONDARY OUTCOMES:
Tinnitus incidence | at inclusion, at 3 weeks, at 6 weeks, 3 months after treatment, 6 months, 12 months and 18 months
  According to Subjective, Objective, Management, Analytic- Late Effects Normal Tissue scales :SOMA-LENT scale (grade 1 to 4).
Hearing loss incidence | at inclusion, at 3 weeks, 6 weeks, 3 months after treatment, 6 months, 12 months and 18 months
  audiogram with measures at 0,25, 0,5, 1, 2, 4, 6, 8, 10 and 12,5 kHz
Association between the onset of tinnitus and/or hearing loss and quality of life | at inclusion, at 3 weeks, 6 weeks, 3 months after treatment, 6 months, 12 months and 18 months
  Evaluation quality of life (Tinnitus Handicap Inventory)
Association between the onset of tinnitus and/or hearing loss and quality of life | at inclusion, at 3 weeks, 6 weeks, 3 months after treatment, 6 months, 12 months and 18 months
  Evaluation quality of life: EVA intensity and discomfort
Association between the onset of tinnitus and/or hearing loss and quality of life | at inclusion, at 3 weeks, 6 weeks, 3 months after treatment, 6 months, 12 months and 18 months
  Evaluation quality of life: EQ-5D-5L questionnaire
Evolution of hearing disorders (tinnitus and/or hearing loss) | at inclusion, at 3 weeks, 6 weeks, 3 months after treatment, 6 months, 12 months and 18 months
  using SOMA-LENT criteria and audiogram
Association between radiotherapy dose received on the cochlea and the onset of tinnitus | 3 months after treatment
  mean dose and max dose
Association between radiotherapy dose received on the cochlea and hearing loss | 3 months after treatment
  mean dose and max dose
Association between cisplatin dose received and the onset of tinnitus and/or hearing loss | 3 months after treatment
  dose in mg/m2
Quality of life after hearing aid fitting in patients requiring hearing aid during/after treatment | at 3 weeks, 6 weeks, 3 months after treatment, 6 months, 12 months and 18 months
  APHAB (Abbreviated Profile of Hearing Aid Benefit) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Florence HUGUET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Radiotherapy Oncology Service TENON Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided